CLINICAL TRIAL: NCT03298828
Title: CD19 Chimeric Antigen Receptor (CAR) and PD-1 Knockout Engineered T Cells for CD19 Positive Malignant B-cell Derived Leukemia and Lymphoma
Brief Title: CD19 CAR and PD-1 Knockout Engineered T Cells for CD19 Positive Malignant B-cell Derived Leukemia and Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Xiaoyun Shang, Principal Investigator, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMMU-CAR-001
Record Dates: First submitted 2017-07-24; First posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Acute Lymphoblastic Leukemia; Burkitt Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CD19 CAR (Experimental): Patients meeting the eligibility criteria will have leukapheresis to isolate the blood immune cells used to manufacture the CD19 CAR T-cells. Patients will receive lymphodepletion with fludarabine and cyclophosphamide prior to infusion of the CD19 CAR T-cells.
  Interventions: Biological: CD19 CAR T-cells
- CD19 CAR and PD-1 knock out (Experimental): Patients meeting the eligibility criteria will have leukapheresis to isolate the blood immune cells used to manufacture the CD19 CAR and PD-1 knock out engineered T-cells. Patients will receive lymphodepletion with fludarabine and cyclophosphamide prior to infusion of the CD19 CAR and PD-1 knock out engineered T-cells.
  Interventions: Biological: CD19 CAR and PD-1 knock out engineered T-cells

INTERVENTIONS:
Biological: CD19 CAR and PD-1 knock out engineered T-cells — A single dose of 1 x 10^6/kg CD19 CAR transduced and PD-1 knock out engineered T-cells will be given as an intravenous injection through a Hickman line or PICC line(peripherally inserted central catheter) on day 0.
  Arms: CD19 CAR and PD-1 knock out
Biological: CD19 CAR T-cells — A single dose of 1 x 10^6/kg CD19 CAR transduced T-cells will be given as an intravenous injection through a Hickman line or PICC line(peripherally inserted central catheter) on day 0.
  Arms: CD19 CAR

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy and blood kinetics of autologous T cells genetically modified to express CD19 Chimeric Antigen Receptor and PD-1 knockout engineered T cells in patients with relapsed or refractory B-Cell Non-Hodgkin Lymphoma and Leukaemia.

DETAILED DESCRIPTION:
This is a multi-centre, non-randomised, open label Phase I clinical trial of an Advanced Therapy Investigational Medicinal Product named CD19 Chimeric Antigen Receptor (CAR) and PD-1 knock out engineered T-cells (CD19 CAR and PD-1 knock out engineered T-cells) in children and adults (age <70 years) with high risk, relapsed CD19+ haematological malignancies (Acute Lymphoblastic Leukemia and Burkitt's lymphoma). Following informed consent and registration to the trial, patients will undergo an unstimulated leukapheresis for the generation of the CD19 CAR T-cells. Patients will receive the CD19 CAR and PD-1 knock out engineered T-cells following lymphodepleting chemotherapy. The study will evaluate the safety, efficacy and duration of response of the CD19 CAR and PD-1 knock out engineered T-cells in children with high risk relapsed CD19+ malignancies.

ELIGIBILITY:
Inclusion Criteria:

* 1.Children and adults (age 70 years or younger) with high risk/relapsed CD19+ haematological malignancy:

  1. Resistant disease (>25% blasts) at end of UKALL 2011 or equivalent induction
  2. ALL with persistent high level MRD at 2nd time point of frontline national protocol (currently > 5 x 10-3 at week 14 UKALL2011 or equivalent)
  3. High risk infant ALL (age < 6 months at diagnosis with MLL gene rearrangement and either presenting white cell count > 300 x 109/L or poor steroid early response (i.e circulating blast count >1x109/L following 7 day steroid pre- phase of Interfant 06)
  4. Intermediate risk infant ALL with MRD > 10-3 at end of Interfant06 induction
  5. Very early (< 18 months from diagnosis) bone marrow or extramedullary relapse of acute lymphoblastic leukaemia (ALL)
  6. Early (within 6 months of finishing therapy) bone marrow, or combined extramedullary relapse of ALL with bone marrow minimal residual disease (MRD) > 10-3 at end of re-induction
  7. Any on therapy relapse of ALL in patients age 16-70
  8. Any relapse of infant ALL
  9. ALL post ≥ 2nd relapse
  10. Any refractory relapse of ALL
  11. ALL with MRD >10-4 prior to planned stem cell transplant
  12. Any relapse of ALL eligible for stem cell transplant but no available HLA matched donor or other contraindication to transplant
  13. Any relapse of ALL after stem cell transplant
  14. Any relapse of Burkitt's or other CD19+ lymphoma
* 2.Agreement to have a pregnancy test, use adequate contraception (if applicable)
* 3.Written informed consent

Exclusion Criteria:

* Exclusion Criteria for registration:

  1. CD19 negative disease
  2. Active hepatitis B, C or HIV infection
  3. Oxygen saturation ≤ 90% on air
  4. Bilirubin > 3 x upper limit of normal
  5. Creatinine > 3 x upper limit of normal
  6. Women who are pregnant or lactating
  7. Stem Cell Transplant patients only: active acute graft-versus-host disease (GVHD) overall Grade ≥ II (Seattle criteria) or moderate/severe chronic GVHD (NIH consensus criteria) requiring systemic steroids
  8. Inability to tolerate leucapheresis
  9. Karnofsky (age ≥ 10 years) or Lansky (age < 10) score ≤ 50%
* Exclusion criteria for CD19CAR T-cell infusion:

  1. Severe intercurrent infection at the time of scheduled CD19 CAR and PD-1 Knockout Engineered T Cells infusion
  2. Requirement for supplementary oxygen or active pulmonary infiltrates at the time of scheduled CD19 CAR and PD-1 Knockout Engineered T Cells infusion
  3. Allogeneic transplant recipients with active acute GVHD overall grade >2 or moderate/severe chronic GVHD requiring systemic steroids at the time of scheduled CD19 CAR and PD-1 Knockout Engineered T Cells infusion

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Molecular remission | 1 month
  Efficacy will be assessed by determining Minimal Residual Disease in the bone marrow aspirate using immunoglobulin heavy chain (IgH) quantitative polymerase chain reaction (qPCR) and/or Next Generation Sequencing in all patients. The proportion of patients achieving molecular remission at 1 month post CD19 CAR and PD-1 Knockout Engineered T-cell infusion will be determined.

SECONDARY OUTCOMES:
Long term molecular remission | 2 years
  Number of patients in molecular remission without further therapy at 2 years
Frequency of circulating CD19 CAR and PD-1 Knockout Engineered T-cells | 2 years
  Persistence and frequency of circulating CD19 CAR and PD-1 Knockout Engineered T-cells in the peripheral blood by flow cytometry and qPCR analyses.
Incidence of hypogammaglobulinaemia | 2 years
  Incidence and duration of hypogammaglobulinaemia.
Relapse rate | 10 years
  Relapse rate monitored during interventional phase and long term follow up for a total of 10 years post cell infusion. Number of patients who relapsed can be summarized as a percentage (for all patients registered to the trial, and also only for those who received the cell infusion).
Overall Survival | 10 years
  Overall survival is monitored during interventional phase and long term follow up for 10 years post-CD19 CAR and PD-1 Knockout Engineered T-cell infusion. Number of patients alive can be summarized as a percentage (for all patients registered to the trial, and also only for those who received the cell infusion).

IPD SHARING:
Plan to Share IPD: Undecided